CLINICAL TRIAL: NCT02738632
Title: Randomized, Double-Blind, Multi-Center, Phase 3 Trial to Evaluate the Efficacy and Safety of Telmisartan/Amlodipine/Hydrochlorothiazide Combination in Comparison With Telmisartan/Amlodipine Combination for Essential Hypertension Patients Not Controlled by Telmisartan/Amlodipine Combination
Brief Title: Efficacy and Safety of TAH Combination in Comparison With Telmisartan/Amlodipine Combination for Essential Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-TAH-301
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-01

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Telmisartan; telmisartan amlodipine combination; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telmisartan/Amlodipine+Hydrochlorothiazide (Experimental): Telmisartan/Amlodipine combination drug and Hydrochlorothiazide
  Interventions: Drug: Telmisartan/Amlodipine+Hydrochlorothiazide
- Telmisartan/Amlodipine (Active Comparator): Telmisartan/Amlodipine combination drug and Placebo for Hydrochlorothiazide
  Interventions: Drug: Telmisartan/Amlodipine; Drug: Placebo for Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan/Amlodipine+Hydrochlorothiazide — Treatment1:Telmisartan/Amlodipine 40/5mg 1 Tab.and Hydrochlorothiazide 12.5mg 1 Tab.QD
  Treatment2: Telmisartan/Amlodipine 40/5mg 2 Tab.and Hydrochlorothiazide 25mg 1 Tab.QD
  Arms: Telmisartan/Amlodipine+Hydrochlorothiazide
Drug: Telmisartan/Amlodipine — Treatment1:Telmisartan/Amlodipine 40/5mg 1 Tab.and Hydrochlorothiazide 12.5mg Placebo 1 Tab.QD
  Treatment2: Telmisartan/Amlodipine 40/5mg 2 Tab.and Hydrochlorothiazide 25mg Placebo 1 Tab.QD
  Arms: Telmisartan/Amlodipine
Drug: Placebo for Hydrochlorothiazide
  Arms: Telmisartan/Amlodipine

SUMMARY:
Randomized, Double-Blind, Multi-Center, Phase 3 Trial to Evaluate the Efficacy and Safety of Telmisartan/Amlodipine/Hydrochlorothiazide Combination in Comparison with Telmisartan/Amlodipine Combination for Essential Hypertension Patients not Controlled by Telmisartan/Amlodipine Combination

ELIGIBILITY:
Inclusion Criteria:

1. 19 years old or above Koreans living in Korea
2. Patients with uncontrolled essential hypertension at screening time(Visit 1)

   * Naïve: 160 mmHg ≤ sitSBP < 200 mmHg
   * Use antihypertensive drugs:140 mmHg ≤ sitSBP < 200 mmHg
3. Patients with uncontrolled hypertension after Telmisartan/Amlodipine 40/5mg treatment for 6 weeks at randomization(Visit 2)

   - 140 mmHg ≤ sitSBP < 200 mmHg
4. Patients who agreed to participate in the trial

Exclusion Criteria:

1. Test results showing the following values at screening time(Visit 1)

   * The change of mean sitSBP ≥ 20 mmHg or sitDBP ≥ 10 mmHg on target arm between 1st and 2nd measurement
   * screening time(Visit 1), time of randomization(Visit 2): sitDBP ≥ 120 mmHg
2. Patients with secondary blood pressure or suspected of secondary blood pressure (for example,aortic coarctation, primary aldosteronism, renal artery stenosis, pheochromocytoma)
3. -Patients with congestive heart failure(NYHA class III~IV)

   * Patients with unstable angina or myocardial infarction or valvular heart disease within 6 months prior to study entry
   * Patients who have severe ventricular tachycardia, atrial fibrillation, atrial flutter or clinically significant arrhythmia
4. Patients who have history of cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months prior to study entry
5. Type I Diabets Mellitus or Type II Diabetes Mellitus with HbA1c > 9%
6. Patients who have history of severe or malignant retinopathy within 6 months prior to study entry
7. Patients who suspected of Renal dysfunction that may affect the absorption, distribution, metabolism or excretion (Serum Creatinine :> 2mg/dL ), gastrointestinal, haematological, liver disease (AST or ALT > 2.5 times of upper limit of normal range)
8. Patients who should be administered antihypertensive drugs other than clinical trial medication(Diuretics, β-blockers, ACE inhibitors, Angiotensin II Receptor Blocker, Calcium Channel Blockers, α-blockers, Renin Inhibitors, Vasodilators)
9. Patients who should be administered medications prohibited for concomitant use during study period
10. Patients who are dependent on drugs or alcohol
11. Patients with surgical and medical disease that may affect the absorption, distribution, metabolism or excretion
12. Patients with hypersensitivity to the components of investigational drug.
13. Patients with hypersensitivity to Sulfonamide
14. Patients with anuria
15. Patients with hypercalcemia, hyponatremia/hypokalemia
16. Patients with Addison's disease
17. Patients who have hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
18. Patients with any chronic or accute inflammation disease needed to chronic inflammation therapy
19. History of malignant tumor including leukemia, lymphoma within 5 years
20. Patients taking other clinical trial drugs within 30 days from the time of visit for screening
21. Pregnancy, breast-feeding, or child-bearing potential Patients
22. Patients who are judged unsuitable to participate in this study by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The change of sitting systolic blood pressure | From baseline at week 8

SECONDARY OUTCOMES:
The change of sitting systolic blood pressure | From baseline at week 2
The change of sitting diastolic blood pressure | From baseline at week 2 and 8
The ratio of subjects who get normalized blood pressure | at week 2 and 8
Response Rate | at week 2 and 8

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung KC, Oh YS, Cha DH, Hong SJ, Won KH, Yoo KD, Rha SW, Ahn YK, Ahn JC, Jang JY, Hong TJ, Cho SK, Park SH, Hyon MS, Nam CW, Chae IH, Yoo BS, Song JM, Jeong JO, Yoon YW, Kim BS, Yang TH, Cho DK, Kim SH, Choi YJ, Ahn JH, Jeon DW, Kim HS. Efficacy and Tolerability of Telmisartan/Amlodipine + Hydrochlorothiazide Versus Telmisartan/Amlodipine Combination Therapy for Essential Hypertension Uncontrolled With Telmisartan/Amlodipine: The Phase III, Multicenter, Randomized, Double-blind TAHYTI Study. Clin Ther. 2018 Jan;40(1):50-63.e3. doi: 10.1016/j.clinthera.2017.11.006. Epub 2017 Dec 14. PMID 29248384